CLINICAL TRIAL: NCT03172364
Title: A Clinical Study to Assess the Cutaneous and Ocular Local Tolerance of Two Cosmetic Facial Cleansers in Healthy Females With Sensitive Skin Under Normal Conditions of Use
Brief Title: To Investigate the Cutaneous and Ocular Local Tolerance of Two Cosmetic Facial Cleanser in Healthy Females With Sensitive Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 207782
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product 1 (Experimental): All the participants in this arm will receive test product 1 (micellar cleanser) at home twice a day (morning and evening) for 21 (±2) days.
  Interventions: Other: Micellar cleanser
- Test product 2 (Experimental): All the participants in this arm will receive test product 2 (micellar foaming cleanser) at home twice a day (morning and evening) for 21 (±2) days.
  Interventions: Other: Micellar foaming cleanser

INTERVENTIONS:
Other: Micellar cleanser — Participants will apply the micellar cleanser topically twice a day (morning and evening). Micellar cleanser will be applied on cotton pad and wiped over the entire face and closed eye to gently cleanse. No need to rub or rinse the micellar cleanser.
  Arms: Test product 1
Other: Micellar foaming cleanser — Participants will use the micellar foaming cleanser topically twice a day (morning and evening). Micellar foaming cleanser will be massaged gently onto wet skin on the face using fingertips. After which participants will rinse thoroughly and pat the skin dry.
  Arms: Test product 2

SUMMARY:
The objective of this clinical study is to assess the cutaneous and ocular local tolerance of two cosmetic facial cleansers in healthy female participants with sensitive skin under normal conditions of use.

DETAILED DESCRIPTION:
This is an assessor blind (dermatologist and ophthalmologist) clinical in use study to determine the local cutaneous and ocular tolerance of two cosmetic facial cleanser products when used as per the intended instructions for use in a population of healthy female participants with clinically assessed sensitive skin.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical (dermatologist or ophthalmologist) examination
* Fitzpatrick phototype I to IV
* Sensitive Skin (as determined by the lactic acid Stinging test)
* Dermatologist score of zero
* Ophthalmologist score of zero
* Dermatologist assessed Dry or Normal/Combination Skin
* Agreement to comply with the procedures and requirements of the study and to attend the scheduled assessment visits
* Frequent use of facial cosmetic make-up, including eye-make-up (5 out of 7 days per week)

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Any history of significant dermatological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes,) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction
* Presence of open sores, pimples, or cysts at the application site
* Active dermatosis (local or disseminated) that might interfere with the results of the study
* Considered immune compromised
* Participants with dermatographism
* Currently using any medication which in the opinion of the investigator, may affect the evaluation of the study product, or place the participant at undue risk
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs, and corticosteroids up to 2 weeks before screening visit and during the study
* Oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit and during the study
* Intention of being vaccinated during the study period or has been vaccinated within 3 weeks of the screening visit
* Currently receiving allergy injections, or received an allergy injection within 7 days prior to Screening visit, or expects to begin injections during study participation
* Previous history of atopy with regards to allergic reactions, irritation or intense discomfort feelings to topical-use products, cosmetics or medication
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit
* Previous participation in this study
* Recent history (within the last 5 years) of alcohol or other substance abuse
* Any participant who, in the judgment of the Investigator, should not participate in the study
* Any participant with corneal ulcers, keratoconus, blepharitis, meibomitis, pterygium, chemosis, moderately or severe hyperemia or other active ocular diseases
* Any skin marks on the face that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles)
* Prisoner or involuntary incarcerated participant
* Participant from an indigenous tribe
* Participant with a qualified dermatologist assessment of oily skin
* An employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 122 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were enrolled from one center in Campinas, Sao Paulo, Brazil.
Pre-assignment Details: A total of 190 participants were screened for the study, out of which 122 participants were enrolled and 68 participants were not eligible to meet study criteria. Out of 122 enrolled participants, 113 were randomized. Out of 77 nonrandomized participants, 73 did not meet the study criteria, 1 had an adverse event (AE), and 3 were lost to follow-up.
Groups:
- Test Product 1: All the participants in this arm received test product 1 (micellar cleanser) at home twice a day (morning and evening) for 21 (±2) days.
- Test Product 2: All the participants in this arm received test product 2 (micellar foaming cleanser) at home twice a day (morning and evening) for 21 (±2) days.
Period: Overall Study
Arm/Group | Test Product 1 | Test Product 2
Started | 55 | 58
Completed | 53 | 57
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product 1 | Test Product 2 | Total
Number analyzed (Participants) | 55 | 58 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (13.54) | 46.9 (12.82) | 46.4 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 58 | 113
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 7 | 5 | 12
  American Indian or Alaskan Native | 0 | 1 | 1
  Asian - Central/South Asian Heritage | 0 | 0 | 0
  Asian - East Asian Heritage | 0 | 0 | 0
  Asian - Japanese Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White - Arabic/North African Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 35 | 46 | 81
  Multiple | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Combined Dermatologist Score
Description: The intensity of any visual signs of irritation was recorded according to Dermal response score: 0=No evidence of irritation, 1=Minimal erythema; barely perceptible, 2=Definite erythema, readily visible; or minimal edema; or minimal popular response, 3=Erythema and papules, 4=Definite edema, 5=Erythema, edema, and papules, 6=Vesicular eruption, and 7=Strong reaction spreading beyond test site. Dermatologist also provided a superficial irritation score if the dermal response score >0. Superficial irritation score was as follow: grade A/score 0=Slight glazed appearance, grade B/score 1=Marked glazing, grade C/score 2=Glazing with peeling and cracking, grade F/score 3=Glazing with fissures, grade G/score 3=Film of dried serous exudate covering all or portion of the patch, and grade H/score 3=Small petechial erosions and/or scabs. The combined score was equal the sum of the dermal response score plus the numerical equivalent of the superficial irritation score. Full range 0-10.
Time Frame: After 21 (+2) days of test product use
Population: Intent to Treat (ITT, N=113) comprised all randomized subjects who had at least 1 cutaneous or ocular assessment following study product application. No inferential statistic were performed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2
Number analyzed (Participants) | 55 | 58
Participants
  At Day 21, Missing | 1 | 1
  At Day 21, score 0 | 51 | 55
  At Day 21, score 1 | 3 | 2

2. Primary Outcome: Frequency of Combined Ophthalmologist Score
Description: Ocular irritation assessed through the observation of the presence of two factors: Lacrimation Intensity and Conjunctiva Involvement. Conjunctiva involvement score are as follow: 0= None - No involvement, 1= Mild - Conjunctivae (palpebral and bulbar) injected above normal with possible chemosis (swelling); no discharge, 2= Moderate - Conjunctivae injected above normal; obvious swelling; possible discharge, and 3= Severe - Conjunctivae more diffuse, deeper crimson red, individual vessels not easily discernible; excessive swelling and/or discharge. Lacrimal intensity score are as follow: 0= None - No lacrimation observed, 1= Mild-Excessive wetness (no distinct tears), 2= Moderate - A few formed tears (contained in orbit), and 3= Severe - Intense tearing (leaving orbit). The combined ophthalmologist score was calculated in the following way: Combined ophthalmologist score = conjunctiva involvement score + lacrimal intensity score. Full range 0-6.
Time Frame: After 21 (+2) days of test product use
Population: ITT (N=113) comprised all randomized subjects who had at least 1 cutaneous or ocular assessment following study product application. No inferential statistic were performed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2
Number analyzed (Participants) | 55 | 58
Participants
  At Day 21, Missing | 1 | 1
  At Day 21, Score 0 | 54 | 57
  At Day 21, Score 1 | 0 | 0

3. Primary Outcome: Frequency of Combined Dermatologist and Ophthalmologist Score
Description: The combined dermatologist and ophthalmologist score was calculated as the sum of the combined dermatologist score (i.e., dermal response score + superficial irritation score) and the combined ophthalmologist score (i.e., conjunctiva involvement score + lacrimal intensity score). No inferential statistic were performed for this endpoint.The full range was from 0 to 13 where lower scores indicated lower dermal irritation.
Time Frame: After 21 (+2) days of test product use
Population: ITT (N=113) comprised all randomized subjects who had at least 1 cutaneous or ocular assessment following study product application.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2
Number analyzed (Participants) | 55 | 58
Participants
  At Day 21, Missing | 1 | 1
  At Day 21, 0 | 51 | 55
  At Day 21, 1 | 3 | 2

4. Primary Outcome: Combined Dermatologist and Ophthalmologist Score (Modified)
Description: A modified combined dermatologist and ophthalmologist score was calculated, where the superficial irritation component was removed from the equation. Therefore, the modified combined dermatologist and ophthalmologist score was defined as the dermal response score + the combined ophthalmologist score (i.e., conjunctiva involvement score + lacrimal intensity score). No inferential statistic were performed for this endpoint.The full range was from 0 to 13 where lower scores indicated lower dermal irritation.
Time Frame: After 21 (+2) days of test product use
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2
Number analyzed (Participants) | 55 | 58
Participants
  At Day 21, Missing | 1 | 1
  At Day 21, 0 | 51 | 55
  At Day 21, 1 | 3 | 2

5. Secondary Outcome: Frequency of Participant Self-assessment Combined Score for Question Responses With Regards to Product Use Experience on Face
Description: Participants asked Subject Self-Assessment questions at Baseline (Visit 2), prior to test product use, 1 hour (± 20 minutes) following first supervised product use, and following 21 (+2) days of product use. Participants scored each symptom asked in the question (Are you experiencing any redness, dryness, burning, itching or stinging of your face?) by using following score: 0= None, 1=Mild, 2= Moderate, and 3= Severe. Combined score face was obtained by summing the 5 subject assessments for face i.e. redness, dryness, burning, itching and stinging. Maximum observed value of this combined score was 3 and maximum possible combined score was 15. Minimum observed value of this combined score was 0 and minimum possible combined score was 0.
Time Frame: Baseline and after 21 (+2) days of test product use
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2
Number analyzed (Participants) | 55 | 58
Participants
  At Baseline, Missing | 0 | 0
  At Baseline, 0=None | 48 | 50
  At Baseline, 1=Mild | 7 | 6
  At Baseline, 2=Moderate | 0 | 2
  At Baseline, 3=Severe | 0 | 0
  At Day 21, Missing | 1 | 1
  At Day 21, 0=None | 48 | 45
  At Day 21, 1=Mild | 6 | 11
  At Day 21, 2=Moderate | 0 | 1
  At Day 21, 3=Severe | 0 | 0

6. Secondary Outcome: Frequency of Participant Self-assessment Combined Score for Question Responses With Regards to Product Use Experience on Eye
Description: Participants asked Subject Self-Assessment questions at Baseline (Visit 2), prior to test product use, 1 hour (± 20 minutes) following first supervised product use, and following 21 (+2) days of product use. Participants scored each symptom asked in the question (Are you experiencing any redness, dryness, burning, itching or stinging of your eyes?) by using following score: 0= None, 1=Mild, 2= Moderate, and 3= Severe. Maximum observed value of this combined score was 3 and maximum possible combined score was 15. Minimum observed value of this combined score was 0 and minimum possible combined score was 0.
Time Frame: Baseline and after 21 (+2) days of test product use
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2
Number analyzed (Participants) | 55 | 58
Participants
  At Baseline, Missing | 0 | 0
  At Baseline, 0 | 55 | 58
  At Baseline, 1 | 0 | 0
  At Baseline, 2 | 0 | 0
  At Baseline, 3 | 0 | 0
  At Day 21, Missing | 1 | 1
  At Day 21, 0 | 54 | 57
  At Day 21, 1 | 0 | 0
  At Day 21, 2 | 0 | 0
  At Day 21, 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 21 days
Arm/Group | Test Product 1 | Test Product 2
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/58
Other Adverse Events (participants affected / at risk) | 5/55 | 4/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product 1 (N=55) | Test Product 2 (N=58)
DRY EYE (Eye disorders) | 1 | 0
OCULAR HYPERAEMIA (Eye disorders) | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 0
ORAL HERPES (Infections and infestations) | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 1
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0
ACNE (Skin and subcutaneous tissue disorders) | 0 | 1
PAPULE (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 1
LIP ULCERATION (Gastrointestinal disorders) | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT03172364/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03172364/SAP_001.pdf